CLINICAL TRIAL: NCT02889913
Title: When Asking the Indication of a Skin Biopsy From a Patient With a Leg Ulcer in Primary Care? Retrospective Study of 100 Consecutive Biopsies
Brief Title: When Asking the Indication of a Skin Biopsy From a Patient With a Leg Ulcer in Primary Care?
Acronym: BIOPULCER
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: Biopsie cutanée
Record Dates: First submitted 2016-08-19; First posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-08

CONDITIONS: Varicose Ulcer; Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention only description — No intervention only description

SUMMARY:
Leg ulcers are frequent. There are no epidemiological studies available in France, but international studies estimate the prevalence between 0.045 and 0.63% of the total population, prevalence increases with age, reaching 5% of patients over 80 years. Extrapolating these prevalences in the French population between 28 000 and 395 000 people are affected in France a leg ulcer.

It is a costly disease. In 2001, a French study conducted among 800 physicians, including 85.7% of general practitioners, involving more than 1000 patients with venous ulcers, it was estimated that the total cost of treatment per patient average was 888 32 euros. This is truly a public health problem.

Leg ulcers are in 80% of cases of vascular causes (venous, arterial or arteriovenous mixed). However, there are rare causes of ulcers: skin carcinoma, infectious ulcers and vasculitis. These ulcers rare causes require specific treatments that can often heal. To diagnose, to perform a skin biopsy. Thus, the general practitioner must know when to put the indication for biopsy of a leg ulcer.

DETAILED DESCRIPTION:
Goal :

Analyzing the last 100 consecutive skin biopsies performed in patients carriers of chronic leg ulcers, followed in the vascular medicine department of the Hospital Saint Joseph Paris, to determine:

* The reasons which motivated the doctor make the indication of biopsy:
* Disease duration of ulcer
* Unusual clinical features
* Other signs associated with ulcer
* Absence of a satisfactory explanation vascular
* The pathological results Purpose: To clear a typical profile ulcers biopsy

Methodology :

* Retrospective, single-center,
* Acquisition of data: via the pathology laboratory of the hospital will be collected the last 100 consecutive biopsies performed with leg ulcers in vascular medicine department of the hospital Saint Joseph Paris, between 1 January 2013 and the October 1, 2013. Then be analyzed all paper and electronic records of these patients.
* Grid and Analysis:

  * Patient histories,
  * vascular profile of patients,
  * clinical and chronological criteria of the ulcer,
  * Other signs associated with ulcer
  * Results of histological biopsies.
* The data will be made anonymous on the grid for collection by a numbering system 1 100.

ELIGIBILITY:
Inclusion Criteria:

* The last 100 consecutive skin biopsies performed in patients carriers of chronic leg ulcers, hospitalized in the vascular medicine department of the Hospital Saint Joseph Paris

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The last 100 consecutive skin biopsies performed in patients carriers of chronic leg ulcers, hospitalized in the vascular medicine department of the Hospital Saint Joseph Paris
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Assessment of disease duration of ulcer | Day 1 of ulceration to the day 30
  by calculating the number of days from ulceration to the healing

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France